CLINICAL TRIAL: NCT01556126
Title: Prove ART (Abluminal Reservoir Technology) Clinical Benefit in Alla Comers Patients
Brief Title: Clinical Performance of CRE8 Drug Eluting Stent in All Comer Population
Acronym: PARTICIPATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CID - Carbostent & Implantable Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C21102
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Stable Angina; Unstable Angina; Acute Myocardial Infarction
Keywords: Coronary artery disease; Drug Eluting Stent; All comers patients
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amphilimus eluting stent (Cre8) (Experimental): Sirolimus formulated coronary eluting stent
  Interventions: Device: Amphilimus Eluting Stent (CRE8)

INTERVENTIONS:
Device: Amphilimus Eluting Stent (CRE8) — Sirolimus formulated coronary eluting stent
  Other Names: CRE8

SUMMARY:
The aim of this study is to evaluate safety and efficacy performances of CRE8 Drug Eluting Stent, in patients comparable to the everyday's clinical practice population, with a specific focus on diabetics, that will be part of a pre-specified study subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients with symptoms of stable angina or documented silent ischemia;
* Patient with coronary artery disease ranging between 0 and 22 according to the Syntax score;
* Patients with acute coronary syndrome, including unstable angina, NSTEMI and STEMI;
* Patient is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for surgical revascularization (CABG);
* Left ventricular ejection fraction > 30%;
* Target de-novo lesions with diameter stenosis > 50% (including total occlusion);
* Target lesion located in a target vessel with a diameter ranging from 2.5 to 4.0 mm;
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Female with childbearing potential or lactating;
* Known allergies to antiplatelets, anticoagulants, contrast media, sirolimus or cobalt chromium;
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.5 mg/dl or on dialysis);
* Thrombocytopenia (platelet count less than 100,000/mm³) or hypercoagulable disorder;
* Known significant gastro-intestinal or urinary bleeding within the past 6 months;
* Patient refusing blood transfusion;
* Patient currently under immunosuppressant therapy;
* Patient with planned surgery within 6 months from the index procedure unless dual antiplatelet therapy is maintained throughout the peri-surgical period;
* Co-morbidities that could interfere with completion of study procedures, or life expectancy less than 1 year;
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study;
* Patient underwent target vessel revascularization with a DES within 3 months prior to the index procedure;
* Target lesion is located or supplied by an arterial or venous bypass graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1191 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical composite endpoint: Cardiac death/Target vessel MI/Clinically indicated TLR | 6 months

SECONDARY OUTCOMES:
Clinical composite endpoints: - Cardiac death/Target vessel MI/Clinically indicated TLR - All death/All MI/All Repeat Revascularization | At 30 days, 1 year and yearly up to 5 years
Stent thrombosis | within 24 hours, 1 month, 6 months, 1 year and yearly up to 5 years
Angiographic in-stent and in-segment endpoints (in the first 100 patients included in the pre-specified diabetic subgroup). | At 6 months
  reference vessel diameter; minimal lumen diameter; % diameter stenosis; binary restenosis; late lumen loss

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — Fondazione San Raffaele del Monte Tabor
Locations (23):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Ziekenhuis Oost Limburg, Genk, Belgium
- Italy (14):
  - Azienda USL 8 Arezzo - Ospedale San Donato, Arezzo, AR
  - A.S.L. CN1 - Ospedale SS Annunziata di Savigliano, Savigliano, CN
  - Istituto Clinico Città Studi, Milan, MI
  - Fondazione San Raffaele del Monte Tabor, Milan, MI
  - Centro Cardiologico Monzino, Milan, MI
  - Istituto Clinico Humanitas IRCCS, Rozzano, MI
  - Azienda di Rilievo Nazionale e di Alta Specializzazione - Presidio Ospedaliero "Civico e Benfratelli", Palermo, PA
  - Azienda Ospedaliera di Padova, Padua, PD
  - Azienda Ospedaliera S. Salvatore, Pesaro, PU
  - Azienda Policlinico Umberto I, Roma, RM
  - Azienda Sanitaria Locale n°2 Savonese - Ospedale San Paolo, Savona, SV
  - ASL TO2 Torino Nord - Ospedale S. Giovanni Bosco, Torino, TO
  - Clinica Mediterranea SpA, Napoli
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
  - TweeSteden Ziekenhuis, Tilburg
- Oslo University Hospital - Rikshospitalet, Oslo, Norway
- Poland (2):
  - Klinika Kardiologii SPSK4 w Lublinie, Lublin
  - Szpital Kliniczny Przemienienia Panskiego, Poznan